CLINICAL TRIAL: NCT06942975
Title: Evaluation of Tuberculosis Treatment Outcomes Before, During and After COVID-19 in a Dedicated Outpatient Unit
Brief Title: Evaluation of Tuberculosis Treatment Outcomes
Acronym: CLIO-TB
Status: Completed | Type: Observational
Sponsor: Azienda Ospedaliera SS. Antonio e Biagio e Cesare Arrigo di Alessandria (Other)
Responsible Party: Sponsor
Other Study IDs: ASO.MInf.23.01
Record Dates: First submitted 2025-04-17; First posted 2025-04-24 (Actual); Last update posted 2025-04-24 (Actual); Status verified 2025-04

CONDITIONS: Tuberculosis
Keywords: Tuberculosis; COVID-19
MeSH Terms: conditions — Tuberculosis; COVID-19

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Other: Patients with turberculosis — The study plans to collect data from patients with microbiological confirmation of tuberculosis, notified to the SS Hospital Infection Surveillance and Control Antimicrobial Stewardship, in the period between 2019 and 2023, taken in charge by the SC Infectious Diseases of the A.O. SS Antonio e Biagio and Cesare Arrigo of Alessandria (Piedmont Region, Italy).

SUMMARY:
Tuberculosis (TB) is an infectious disease caused by Mycobacterium species grouped in the Mycobacterium tuberculosis complex. TB remains a major global health problem, despite the fact that there are drugs that can eradicate the infection. The study aims to describe the clinical, microbiological, therapeutic and prognostic characteristics of TB patients afferent to the SC Infectious Diseases of A.O. SS Antonio e Biagio e Cesare Arrigo of Alexandria during 2019-2022 and, secondarily, to evaluate the treatment outcomes (as defined by the World Health Organization) of TB patients afferent to the SC Infectious Diseases of A. O. SS Antonio e Biagio e Cesare Arrigo of Alexandria considering the influence of the SARS-CoV-2 pandemic (pre-pandemic, inter-pandemic and post-pandemic period) and to evaluate the post-treatment relapse rate.

DETAILED DESCRIPTION:
Tuberculosis (TB) is an infectious disease caused by Mycobacterium species grouped in the Mycobacterium tuberculosis complex. TB remains a major global health problem, despite the fact that there are drugs that can eradicate the infection. Of concern, however, are both underdiagnosis and the circulation of strains resistant to first-line therapies. Indeed, if not properly administered, TB treatment regimens are associated with unfavorable outcomes, promoting the circulation of the bacterium and the emergence of drug resistance. Monitoring the effectiveness of tuberculosis treatment is therefore of paramount importance in both clinical practice and surveillance to maximize the quality of individual patient care and the effectiveness of public health actions. The COVID-19 pandemic has created unprecedented challenges for populations, public health departments, and health facilities worldwide, and is likely to have devastating effects on global TB prevention and control programs, including a reversal of the progress achieved over the past decade.The present study aims to describe the case history of TB patients afferent to A.O. SS Antonio e Biagio and Cesare Arrigo in Alexandria and to evaluate treatment outcomes. This facility underwent a disruption of services during the pandemic period, and also initiated in the post-pandemic period a TB clinical management service with an active retention-in-care approach, generating appointments for follow-up visits and contacting patients who did not keep these appointments.

ELIGIBILITY:
Inclusion Criteria:

* Patients aged ≥18 years
* Patients with tuberculosis with microbiological confirmation
* Patients notified to the SS Surveillance and Control Hospital Infections Antimicrobial Stewardship of the Alexandria Hospital Company from 2019 to 2023
* Patients taken in charge by the SC Infectious Diseases of the Alexandria Hospital Company for whom MOD B has been completed
* Obtaining informed consent

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: The study plans to enroll patients with microbiological confirmation of tuberculosis, notified to the SS Surveillance and Control of Hospital Infections Antimicrobial Stewardship, during the period between 2019 and 2022, taken over by the Infectious Diseases SC of the A.O. SS Antonio e Biagio and Cesare Arrigo of Alessandria, Italy.
Sampling Method: Probability Sample
Enrollment: 111 (Actual)
Dates: Start 2023-05-08 (Actual); Primary Completion 2023-11-09 (Actual); Study Completion 2023-12-12 (Actual)

PRIMARY OUTCOMES:
Description of patient characteristics | Baseline
  Description of the characteristics of TB patients referred to the SC Infectious Diseases of the A.O. SS Antonio e Biagio and Cesare Arrigo of Alexandria in the period 2019-2023

SECONDARY OUTCOMES:
Number of cured patients | Baseline
  Number of patients treated at the SC Infectious Diseases who are "cured" as a treatment outcome
Number of deceased patients | Baseline
  Number of patients treated at the SC Infectious Diseases who are "dead" as a treatment outcome
Number of patients lost to follow-up | Baseline
  Number of patients treated at the SC Infectious Diseases who are "lost to follow-up" as a treatment outcome
Number of post-treatment relapses | Baseline
  Number of post-treatment relapses

CONTACTS AND LOCATIONS:
Locations (1):
- Clinical Trial Center, Alessandria, Italy, Italy

IPD SHARING:
Plan to Share IPD: No